CLINICAL TRIAL: NCT00593385
Title: Atrium iCAST Iliac Stent Pivotal Study
Acronym: iCARUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Atrium Medical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Atrium 701
Record Dates: First submitted 2008-01-02; First posted 2008-01-15 (Estimated); Results first posted 2018-05-17 (Actual); Last update posted 2018-05-17 (Actual); Status verified 2018-04

CONDITIONS: Peripheral Vascular Disease
Keywords: Symptomatic claudication or rest pain and angiographic confirmation of either de novo or restenotic lesions in the common and/or external iliac artery.
MeSH Terms: conditions — Peripheral Vascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- iCAST covered stent (Other): This is a one arm trial. All subjects received the iCAST covered stent.
  Interventions: Device: iCAST covered stent

INTERVENTIONS:
Device: iCAST covered stent — Iliac stent implantation

SUMMARY:
Prospective, multicenter, non-randomized, single-arm registry to evaluate the safety and effectiveness of the iCAST Covered Stent System in the treatment of patients with symptomatic claudication or rest pain and angiographic confirmation of de novo or restenotic lesions in the common and/or external iliac artery.

DETAILED DESCRIPTION:
STUDY DESIGN: Prospective, multicenter, non-randomized, single-arm registry

OBJECTIVE: The primary objective is to evaluate the iCAST covered stent to a performance metric derived from studies of FDA-approved iliac stent devices for treating iliac artery stenoses in patients with de novo or restenotic lesions in the common and/or external iliac arteries.

NUMBER OF SUBJECTS: 165 subjects, including up to 25 subjects with totally occluded lesions.

PRIMARY ENDPOINTS: The primary endpoint is a composite endpoint defined as the occurrence of death within 30 days, target site revascularization or restenosis (by ultrasound determination) within 9 months post-procedure.

SECONDARY ENDPOINTS: Secondary endpoints include:

1. Major adverse vascular events (MAVE) defined as a composite rate of myocardial infarction at 30 days, stent thrombosis, clinically apparent distal embolization, defined as causing end-organ damage (e.g. lower extremity ulceration, tissue necrosis, or gangrene), arterial rupture, acute limb ischemia, target limb amputation or procedure related bleeding event requiring transfusion.
2. A major adverse event (MAE) is defined as a composite rate of MAVE or any death, or stroke, up to 30 days post-procedure.
3. Device success, defined as the successful delivery and deployment of the study stent and intact retrieval of the delivery system.
4. Acute procedural success, defined as device success and achievement of < 30% residual stenosis immediately after stent deployment, mean transtenotic pressure gradient of < 5 mmHg and without occurrence of in-hospital MAVE.
5. Clinical success, assessed both early (30 days) and late (6, 9 and 12 months).
6. Patency assessed at each follow-up time point, categorized as primary, primary-assisted or secondary patency.
7. Composite rate of 30 day death, 9 month target site revascularization and 9 month restenosis in subjects without iliac total occlusions.

PATIENT POPULATION: Eligible patients have symptomatic claudication or rest pain and angiographic confirmation of either de novo or restenotic lesions in the common and/or external iliac artery.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is 18 years of age or older.
2. Subject has lifestyle limiting claudication or rest pain (Rutherford-Becker scale 2-4).
3. Presence of de novo and/or restenotic lesions in the common and/or external iliac artery.
4. Subject has single, bilateral or multiple target lesions that is (are) ≥ 50% stenosed by visual estimate.
5. The target lesion(s) can be successfully crossed with a guide wire and dilated.
6. The target segment of subject's lesion(s) is between 5 and 12mm in diameter and less than 110 mm in length.
7. Subject has angiographic evidence of a patent profunda or superficial femoral artery (SFA) in the target limb.
8. Subject has provided written informed consent.
9. Subject is able and willing to adhere to the required follow-up visits and testing through month 36.
10. Subject is able and willing to adhere to the required follow-up medication regimen.

Exclusion Criteria:

1. Presence of other non-target ipsilateral arterial lesions requiring treatment within 30 days post-procedure (Note that treatment of ipsilateral SFA lesions may be allowed under certain circumstances). Treatment of lesions in any other vascular bed must be completed at least 30 days prior to enrollment.
2. The target lesion(s) has adjacent, acute thrombus.
3. The target lesion(s) is highly calcified or was previously treated with a stent.
4. Target lesion involves the internal iliac artery resulting in crossing of the side-branch with the iCAST device (e.g. "jailing" of the side-branch).
5. Subject has an abdominal aortic aneurysm contiguous with the iliac artery target lesion.
6. Subject has a pre-existing target iliac artery aneurysm or perforation or dissection of the target iliac artery prior to initiation of the iCAST implant procedure.
7. Subject has a post-surgical stenosis and anastomotic suture treatments of the target vessel.
8. Subject has a vascular graft previously implanted in the native iliac vessel.
9. Subject has tissue loss, defined as Rutherford-Becker classification category 5 or 6.
10. Subject has contrast agent hypersensitivity that cannot be adequately pre-medicated, has a hypersensitivity to stainless steel, expanded polytetrafluoroethylene (ePTFE) or has intolerance to antiplatelet, anticoagulant, or thrombolytic medications.
11. History of neutropenia (WBC <3,000/mm3), coagulopathy, or thrombocytopenia (platelet count <80,000/ μL) that has not resolved or has required treatment in the past 6 months.
12. Known bleeding or hypercoagulability disorder or significant anemia (Hb< 8.0) that cannot be corrected.
13. Subject has the following laboratory values:

    1. platelet count less than 80,000/ μL,
    2. prothrombin time (PT)/partial thromboplastin time (PTT) not within normal limits
    3. serum creatinine level greater than 2.5 mg/dL
14. Subject requires general anesthesia for the procedure.
15. Subject is pregnant.
16. Subject has a co-morbid illness that may result in a life expectancy of less than 1 year.
17. Subject is participating in an investigational study of a new drug, biologic or device at the time of study screening. Note: Subjects who are participating in the long term follow-up phase of a previously investigational and now FDA-approved product are not excluded by this criterion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2007-10; Primary Completion 2011-08 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John R Laird, MD, Principal Investigator — Adventist Health
Locations (25):
- United States (24):
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Fogarty Clincal Research Incorporated, Mountain View, California
  - University of California, Davis, Sacramento, California
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Piedmont Hospital Research Institute, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Krannert Institute of Cardiology, Indianapolis, Indiana
  - University of Louisville, Louisville, Kentucky
  - Terrebonne General Medical Center, Houma, Louisiana
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Mass General Hospital, Boston, Massachusetts
  - Forest General Hospital, Hattiesburg, Mississippi
  - Kansas City Heart Foundation, Kansas City, Missouri
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Duke University Medical Center, Durham, North Carolina
  - Lindner Clinical Trial Center, Cincinnati, Ohio
  - University Hospitals, Case Medical Center, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - MidWest Cardiology Research Foundation, Columbus, Ohio
  - Holy Spirit Cardiovascular Institute, Camp Hill, Pennsylvania
  - North Central Heart Institute, Sioux Falls, South Dakota
  - Tennova Healthcare - Turkey Creek Medical Center, Knoxville, Tennessee
  - Cardiovascular Research Institute of Dallas, Dallas, Texas
  - The Methodist Hospital, Houston, Texas
- Herzzentrum Bad Krozingen, Bad Krozingen, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Laird JR, Loja M, Zeller T, Niazi KAK, Foster MT, Ansel G, Stone DH, Dave RM, Popma JJ, Jaff MR, Massaro JM. iCAST Balloon-Expandable Covered Stent for Iliac Artery Lesions: 3-Year Results from the iCARUS Multicenter Study. J Vasc Interv Radiol. 2019 Jun;30(6):822-829.e4. doi: 10.1016/j.jvir.2018.12.707. Epub 2019 Apr 25. PMID 31031089

RESULTS

PARTICIPANT FLOW:
Groups:
- Device: ICAST Covered Stent: Implantation of ≥ 1 ICAST stent
Period: Overall Study
Arm/Group | Device: ICAST Covered Stent
Started | 165
Intention to Treat (ITT) Population (Subjects who signed written informed consent, enrolled in the study and met study entry criteria.) | 152 (Excludes 13 subjects who did not meet inclusion/exclusion criteria.)
Completed | 125 (125 of 165 enrolled patients completed the study.)
Not Completed | 40
Not completed — Death | 14
Not completed — Lost to Follow-up | 17
Not completed — Withdrawal by Subject | 9

BASELINE CHARACTERISTICS:
Population: ITT population was assessed for baseline measures: this includes subjects who signed the written informed consent, enrolled in the study and met the study entry criteria.
Arm/Group | Device: ICAST Covered Stent
Number analyzed (Participants) | 152
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.23 (9.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58
  Male | 94
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 149
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 8
  White | 142
  More than one race | 2
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 132
  Germany | 20
Cigarette Smoking Status [Count of Participants; unit: Participants] — Population: One subject was missing data.
  Participants
    number analyzed (Participants) | 151
    Current smoker | 76
    Former smoker | 62
    Non-smoker | 13
    Unknown | 0
Previous Peripheral Artery Revascularization/Surgery [Count of Participants; unit: Participants] — Population: Two subjects were missing data.
  Participants
    number analyzed (Participants) | 150
    (all) | 25
Coronary Artery Disease [Count of Participants; unit: Participants] — Population: One subject was missing data.
  Participants
    number analyzed (Participants) | 151
    (all) | 77
Previous Myocardial Infarction (MI) [Count of Participants; unit: Participants] — Population: One subject was missing data.
  Participants
    number analyzed (Participants) | 151
    (all) | 35
Previous percutaneous coronary revascularization [Count of Participants; unit: Participants] — Population: One subject was missing data.
  Participants
    number analyzed (Participants) | 151
    (all) | 39
Coronary Artery Bypass Graft Surgery [Count of Participants; unit: Participants] — Population: One subject was missing data.
  Participants
    number analyzed (Participants) | 151
    (all) | 34
Cerebrovascular Accident [Count of Participants; unit: Participants] | 11
Previous Amputation [Count of Participants; unit: Participants] | 2
Transient Ischemic Attack [Count of Participants; unit: Participants] — Population: One subject was missing data.
  Participants
    number analyzed (Participants) | 151
    (all) | 7
Diabetes Mellitus [Count of Participants; unit: Participants] | 56
Hypertension [Count of Participants; unit: Participants] | 129
Hypercholesterolemia [Count of Participants; unit: Participants] | 130
Renal Insufficiency [Count of Participants; unit: Participants] | 19

OUTCOME MEASURES:

1. Primary Outcome: Percentage of ITT Population Experiencing Death Within 30 Days, Target Site Revascularization or Restenosis
Description: The primary endpoint is a composite endpoint defined as the occurrence of death within 30 days, target site revascularization within 9 months or restenosis (by ultrasound determination) at 9 months.
Time Frame: Within 9 Months post-procedure
Population: ITT population: Subjects who signed the written informed consent, enrolled in the study and met the study entry criteria.
Measure: Number; unit: Percentage of subjects
Groups:
- iCAST Covered Stent: Device: iCAST covered stent
  Implantation of ≥1 iCAST stents
Arm/Group | iCAST Covered Stent
Number analyzed (Participants) | 152
Percentage of subjects | 8.1
Statistical Analysis 1: Comparison: iCAST Covered Stent; The composite event rate to determine the performance metric of 16.57% was based on a meta-analysis performed on data from 3 previous studies(9.67%). A 6.9% margin was deemed acceptable at the time of study design. Rejection of the null hypothesis requires that the iCAST Covered Stent primary endpoint rate was significantly below 16.57%. Other assumptions for the analysis included a power of 80% and one-sided alpha error of 5%; Test type: Other; p = 0.005, Exact test of the binomial distribution — An exact one sided upper 95% confidence interval of the primary endpoint rate was calculated based on primary analysis population; Meta-Analysis = 9.67, 95% CI 1-sided [upper limit 16.57] — To estimate primary endpoint rate, a meta-analysis was performed on data from 3 previous studies. The meta-analytical rate derived was 9.67%

2. Secondary Outcome: Acute Procedural Success
Description: Device success and achievement of < 30% residual stenosis immediately after stent placement and without occurrence of in-hospital MAVE.
Time Frame: Post-procedure
Population: Subset of ITT population with available data for analysis (ITT population included subjects who signed the written informed consent, enrolled in the study and met the study entry criteria).
Measure: Count of Participants; unit: Participants
Arm/Group | Device: ICAST Covered Stent
Number analyzed (Participants) | 151
Participants | 140

3. Secondary Outcome: Device Success
Description: Successful delivery and deployment of the study stent and intact retrieval of the delivery system.
Time Frame: Post-procedure
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Device: ICAST Covered Stent
Number analyzed (Participants) | 152
Participants | 150

4. Secondary Outcome: Major Adverse Event (MAE)
Description: Composite rate of MAVE or any death, or stroke.
Time Frame: 30 Days
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Device: ICAST Covered Stent
Number analyzed (Participants) | 151
Participants | 8

5. Secondary Outcome: Major Adverse Vascular Event (MAVE)
Description: Composite rate of myocardial infarction at 30 days, stent thrombosis, clinically apparent distal embolization, arterial rupture, acute limb ischemia, target limb amputation, or procedure related bleeding event requiring transfusion.
Time Frame: 30 Days
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Device: ICAST Covered Stent
Number analyzed (Participants) | 151
Participants | 7

6. Secondary Outcome: Major Adverse Vascular Event (MAVE)
Description: as for outcome 5
Time Frame: 180 Days
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Device: ICAST Covered Stent
Number analyzed (Participants) | 144
Participants | 10

7. Secondary Outcome: Major Adverse Vascular Event (MAVE)
Description: as for outcome 5
Time Frame: 270 Days
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Device: ICAST Covered Stent
Number analyzed (Participants) | 140
Participants | 10

8. Secondary Outcome: Major Adverse Vascular Event (MAVE)
Description: as for outcome 5
Time Frame: 360 Days
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Device: ICAST Covered Stent
Number analyzed (Participants) | 139
Participants | 10

9. Secondary Outcome: Early Clinical Success
Description: Improvement of the Rutherford-Becker clinical criteria by ≥ 1 category. (Classification system for evaluating clinical improvement as defined by Rutherford R, Becker G. Standards for evaluating and reporting the results of surgical and percutaneous therapy for peripheral arterial disease. Journal of Vascular Interventional Radiology 1991;2:169-174.)
Time Frame: 1 Month
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Device: ICAST Covered Stent
Number analyzed (Participants) | 150
Participants | 133

10. Secondary Outcome: Late Clinical Success
Description: Maintained improvement in ankle brachial index (ABI), the ratio of the blood pressure at the ankle to the blood pressure in the upper arm.
Time Frame: 6 Months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Device: ICAST Covered Stent
Number analyzed (Participants) | 126
Participants | 80

11. Secondary Outcome: Late Clinical Success
Description: as for outcome 10
Time Frame: 9 Months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Device: ICAST Covered Stent
Number analyzed (Participants) | 128
Participants | 98

12. Secondary Outcome: Late Clinical Success
Description: as for outcome 10
Time Frame: 12 Months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Device: ICAST Covered Stent
Number analyzed (Participants) | 128
Participants | 86

13. Secondary Outcome: Late Clinical Success
Description: as for outcome 10
Time Frame: 24 Months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Device: ICAST Covered Stent
Number analyzed (Participants) | 113
Participants | 80

14. Secondary Outcome: Late Clinical Success
Description: as for outcome 10
Time Frame: 36 Months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Device: ICAST Covered Stent
Number analyzed (Participants) | 105
Participants | 76

15. Secondary Outcome: Primary Patency
Description: Continuous flow without revascularization, bypass or target limb amputation.
Time Frame: 1 Month
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Device: ICAST Covered Stent
Number analyzed (Participants) | 151
Participants | 151

16. Secondary Outcome: Primary Patency
Description: Continuous flow without revascularization, bypass or target limb amputation.
Time Frame: 6 Months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Device: ICAST Covered Stent
Number analyzed (Participants) | 144
Participants | 143

17. Secondary Outcome: Primary Patency
Description: Continuous flow without revascularization, bypass or target limb amputation.
Time Frame: 9 Months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Device: ICAST Covered Stent
Number analyzed (Participants) | 139
Participants | 134

18. Secondary Outcome: Primary Patency
Description: Continuous flow without revascularization, bypass or target limb amputation.
Time Frame: 12 Months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Device: ICAST Covered Stent
Number analyzed (Participants) | 138
Participants | 129

19. Secondary Outcome: Primary Patency
Description: Continuous flow without revascularization, bypass or target limb amputation.
Time Frame: 24 Months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Device: ICAST Covered Stent
Number analyzed (Participants) | 129
Participants | 113

20. Secondary Outcome: Primary Patency
Description: Continuous flow without revascularization, bypass or target limb amputation.
Time Frame: 36 Months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Device: ICAST Covered Stent
Number analyzed (Participants) | 118
Participants | 100

21. Secondary Outcome: Primary-Assisted Patency
Description: Continuous flow assisted when the target vessel has restenosed at any time post-procedure.
Time Frame: 1 Month
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Groups:
- Device: ICAST Covered Stent: Implantation of ≥1 ICAST stent
Arm/Group | Device: ICAST Covered Stent
Number analyzed (Participants) | 151
Participants | 151

22. Secondary Outcome: Primary-Assisted Patency
Description: Continuous flow assisted when the target vessel has restenosed at any time post-procedure.
Time Frame: 6 Months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Device: ICAST Covered Stent
Number analyzed (Participants) | 144
Participants | 144

23. Secondary Outcome: Primary-Assisted Patency
Description: Continuous flow assisted when the target vessel has restenosed at any time post-procedure.
Time Frame: 9 Months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Device: ICAST Covered Stent
Number analyzed (Participants) | 139
Participants | 139

24. Secondary Outcome: Primary-Assisted Patency
Description: Continuous flow assisted when the target vessel has restenosed at any time post-procedure.
Time Frame: 12 Months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Device: ICAST Covered Stent
Number analyzed (Participants) | 138
Participants | 138

25. Secondary Outcome: Primary-Assisted Patency
Description: Continuous flow assisted when the target vessel has restenosed at any time post-procedure.
Time Frame: 24 Months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Device: ICAST Covered Stent
Number analyzed (Participants) | 129
Participants | 128

26. Secondary Outcome: Primary-Assisted Patency
Description: Continuous flow assisted when the target vessel has restenosed at any time post-procedure.
Time Frame: 36 Months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Device: ICAST Covered Stent
Number analyzed (Participants) | 115
Participants | 114

27. Secondary Outcome: Secondary Patency
Description: Re-establishment of flow to distal arteries after occlusion has occurred at the target vessel.
Time Frame: 1 Month
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Device: ICAST Covered Stent
Number analyzed (Participants) | 151
Participants | 151

28. Secondary Outcome: Secondary Patency
Description: Re-establishment of flow to distal arteries after occlusion has occurred at the target vessel.
Time Frame: 6 Months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Device: ICAST Covered Stent
Number analyzed (Participants) | 144
Participants | 144

29. Secondary Outcome: Secondary Patency
Description: Re-establishment of flow to distal arteries after occlusion has occurred at the target vessel.
Time Frame: 9 Months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Device: ICAST Covered Stent
Number analyzed (Participants) | 139
Participants | 139

30. Secondary Outcome: Secondary Patency
Description: Re-establishment of flow to distal arteries after occlusion has occurred at the target vessel.
Time Frame: 12 Months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Device: ICAST Covered Stent
Number analyzed (Participants) | 138
Participants | 138

31. Secondary Outcome: Secondary Patency
Description: Re-establishment of flow to distal arteries after occlusion has occurred at the target vessel.
Time Frame: 24 Months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Device: ICAST Covered Stent
Number analyzed (Participants) | 129
Participants | 129

32. Secondary Outcome: Secondary Patency
Description: Re-establishment of flow to distal arteries after occlusion has occurred at the target vessel.
Time Frame: 36 Months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Device: ICAST Covered Stent
Number analyzed (Participants) | 115
Participants | 115

ADVERSE EVENTS:
Time Frame: 1080 Days post-procedure
Description: Subjects were encouraged to report AEs spontaneously or in response to general, non-directed questioning.
Arm/Group | Device: ICAST Covered Stent
All-Cause Mortality (participants affected / at risk) | 14/165
Serious Adverse Events (participants affected / at risk) | 86/165
Other Adverse Events (participants affected / at risk) | 22/165
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Device: ICAST Covered Stent (N=165)
Anaemia (Blood and lymphatic system disorders) | 2 (2)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 6 (8)
Angina pectoris (Cardiac disorders) | 3 (5)
Angina unstable (Cardiac disorders) | 3 (4)
Atrial fibrillation (Cardiac disorders) | 2 (2)
Atrial flutter (Cardiac disorders) | 1 (1)
Atrioventricular block (Cardiac disorders) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 7 (9)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1)
Coronary artery disease (Cardiac disorders) | 2 (2)
Coronary artery occlusion (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 6 (6)
Stress cardiomyopathy (Cardiac disorders) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 (4)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Intestinal perforation (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (8)
Pancreatitis acute (Gastrointestinal disorders) | 1 (3)
Peritonitis (Gastrointestinal disorders) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Asthenia (General disorders) | 1 (1)
Catheter site haematoma (General disorders) | 3 (3)
Chest pain (General disorders) | 4 (5)
Impaired healing (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Hepatic steatosis (Hepatobiliary disorders) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 2 (2)
Abdominal abscess (Infections and infestations) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
Bronchitis bacterial (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (1)
Groin abscess (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 8 (11)
Pneumonia staphylococcal (Infections and infestations) | 1 (1)
Post procedural sepsis (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 3 (3)
Urosepsis (Infections and infestations) | 1 (1)
Abdominal wound dehiscence (Injury, poisoning and procedural complications) | 1 (2)
Anaemia postoperative (Injury, poisoning and procedural complications) | 1 (1)
Aortic injury (Injury, poisoning and procedural complications) | 1 (1)
Arterial injury (Injury, poisoning and procedural complications) | 1 (1)
Device dislocation (Injury, poisoning and procedural complications) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1)
In-stent arterial restenosis (Injury, poisoning and procedural complications) | 6 (8)
Incisional hernia (Injury, poisoning and procedural complications) | 1 (1)
Postoperative ileus (Injury, poisoning and procedural complications) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1)
Stent occlusion (Injury, poisoning and procedural complications) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1)
Tendon injury (Injury, poisoning and procedural complications) | 1 (1)
Traumatic brain injury (Injury, poisoning and procedural complications) | 2 (2)
Urostomy complication (Injury, poisoning and procedural complications) | 1 (1)
Vascular graft occlusion (Injury, poisoning and procedural complications) | 2 (2)
Acidosis (Metabolism and nutrition disorders) | 1 (1)
Fluid overload (Metabolism and nutrition disorders) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1)
Obesity (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Fistula (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 2 (2)
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Colon cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Brain mass (Nervous system disorders) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 2 (2)
Cerebrovascular accident (Nervous system disorders) | 3 (3)
Encephalopathy (Nervous system disorders) | 1 (1)
Polyneuropathy (Nervous system disorders) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 2 (2)
Syncope (Nervous system disorders) | 3 (3)
Syncope vasovagal (Nervous system disorders) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 2 (2)
Depression (Psychiatric disorders) | 1 (1)
Calculus ureteric (Renal and urinary disorders) | 1 (1)
Renal artery occlusion (Renal and urinary disorders) | 1 (1)
Renal artery stenosis (Renal and urinary disorders) | 2 (2)
Renal disorder (Renal and urinary disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 5 (5)
Renal failure chronic (Renal and urinary disorders) | 1 (1)
Renal mass (Renal and urinary disorders) | 2 (2)
Galactorrhoea (Reproductive system and breast disorders) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (3)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Psoriasis (Skin and subcutaneous tissue disorders) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Aortic stenosis (Vascular disorders) | 1 (1)
Arterial restenosis (Vascular disorders) | 2 (2)
Arterial thrombosis limb (Vascular disorders) | 1 (1)
Femoral arterial stenosis (Vascular disorders) | 5 (5)
Femoral artery occlusion (Vascular disorders) | 5 (9)
Haemorrhage (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 4 (4)
Iliac artery stenosis (Vascular disorders) | 7 (9)
Intermittent claudication (Vascular disorders) | 7 (9)
Orthostatic hypotension (Vascular disorders) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 5 (5)
Peripheral artery aneurysm (Vascular disorders) | 1 (1)
Peripheral ischaemia (Vascular disorders) | 2 (5)
Peripheral vascular disorder (Vascular disorders) | 1 (1)
Subclavian artery stenosis (Vascular disorders) | 1 (1)
Vascular pseudoaneurysm (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5.0% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Device: ICAST Covered Stent (N=165)
Peripheral artery dissection (Vascular disorders) | 22 (22)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No publication or publicizing of data or results without the Sponsor's prior written permission. Party wishing to publish or publicize will submit proposed manuscript or publication to Sponsor for comment at least 60 days prior to release. Publishing party will make every reasonable attempt to incorporate comments received from Sponsor during 60 day period.The publishing party won't use Sponsor's confidential information in manuscript or publication without the prior written consent of sponsor.